CLINICAL TRIAL: NCT03569475
Title: A Double-blind, Placebo- and Active-controlled Evaluation of the Safety and Efficacy of Levomilnacipran ER in Pediatric Patients 7-17 Years With Major Depressive Disorder
Brief Title: Efficacy, Safety, and Tolerability of Levomilnacipran ER in Pediatric Patients (7-17 Years) With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVM-MD-14
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Levomilnacipran; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Levomilnacipran ER 40-80 mg/day (Experimental): Levomilnacipran extended release (ER) capsules, orally, 10 milligram per day (mg/day) on Days 1 to 3, 20 mg/day on Days 4 to 7, and 40 mg/day from Week 2 through Week 8 of the Double-blind Treatment Period followed by levomilnacipran ER 40 mg/day on Days 1 and 2, and then 20 mg/day from Day 3 through Day 7 in the Down-taper Period. Based on therapeutic response and tolerability, an additional dose increase to 80 mg/day was permitted at Week 3 of the Double-blind Treatment Period.
  Interventions: Drug: Levomilnacipran ER
- Fluoxetine 20 mg/day (Active Comparator): Fluoxetine capsule, orally, 10 mg/day at Week 1, and 20 mg/day from Week 2 through Week 8 of the Double-blind Treatment Period followed by fluoxetine 10 mg/day from Day 1 through Day 7 of the Down-taper Period.
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Matching placebo capsules once daily through 8 weeks in the Double-blind Treatment Period and Days 1 through 7 in the Down-taper Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levomilnacipran ER — Levomilnacipran extended-release oral capsules
  Arms: Levomilnacipran ER 40-80 mg/day
Drug: Fluoxetine — Fluoxetine oral capsules
  Arms: Fluoxetine 20 mg/day
Drug: Placebo — Matching placebo oral capsules
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of levomilnacipran compared with placebo in pediatric outpatients (7-17 years) with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet Diagnostic and statistical manual of mental disorders fifth edition (DSM-5) criteria for MDD, confirmed by Kiddie Schedule for Affective Disorders - Present and Lifetime (K-SADS-PL)
* Patients must have a score ≥ 40 on the Children's Depression Rating Scale-Revised (CDRS-R) at Visits 1 and 2
* Patients must have a Clinical Global Impressions-Severity (CGI-S) score ≥ 4 at Visits 1 and 2
* Patients must have a caregiver who can and is willing to consent to be responsible for safety monitoring of the Patient, provide information about the patient's condition, oversee the administration of investigational product, and accompany the patients to all study visits
* Female patients of childbearing potential who are sexually active must agree to use a reliable method of contraception that will continue for the duration of the study and within 30 days following the end of study participation.
* A sexually active male patients must agree to use contraception as detailed below during the treatment period and for at least 30 days after the last dose of investigational product.

Exclusion Criteria:

* DSM-5-based diagnosis of an axis I disorder other than MDD that is the primary focus of treatment.
* Prior diagnosis of mental retardation or amnestic or other cognitive disorders based on DSM-5 criteria
* Imminent risk of injuring self or others or causing damage to property as judged by the Investigator
* Suicide risk as determined by meeting either of the following criteria:

  * Any suicide attempt within the past year
  * Significant risk at Visit 1 (Screening) or Visit 2 (Baseline), as judged by the Investigator based on the psychiatric interview or information collected in the Columbia-Suicide Severity Rating Scale (C-SSRS) treatment-Related Criteria
* History of allergy, intolerance, or hypersensitivity to levomilnacipran, milnacipran, fluoxetine, or any other Selective serotonin reuptake inhibitors (SSRI) or Serotonin and norepinephrine reuptake inhibitors (SNRI) or known hypersensitivity to the investigational products' non-medicinal ingredients including gelatin and cellulose
* Patients requiring prohibited concomitant medication or herbal supplements that could not be discontinued or switched to an allowable alternative medication and stabilized for at least 2 weeks preceding Visit 2 (Baseline)
* Patients taking any psychoactive drug or psychoactive herbal remedy within 5 half-lives before Baseline (Visit 2), Patients who have ever been treated with a depot antipsychotic must also be excluded
* Patients who have initiated or terminated psychotherapy or behavior therapy within1 month before Visit 1 (Screening), or who plan to initiate or change such therapies during the course of the study Other Medical criteria
* A clinically significant disease state that, in the investigator's opinion, might indicate that the patients is unsuitable for the study
* Any cardiovascular disease or condition that is clinically significant, unstable, or decompensated.
* Hypo- or hyperthyroidism, unless stabilized on appropriate pharmacotherapy with no change in dosage for at least 3 months before Visit 1 (Screening)
* Any condition that would be expected to affect drug absorption (eg, gastric bypass surgery)
* History of seizure disorder (except simple childhood febrile seizures before age 5), unexplained syncope or black-out episodes, stroke, significant head injury, tumor of the central nervous system, or any other condition that predisposes the patient toward a risk for seizure
* History of drug or alcohol abuse or dependence within the past year
* Pregnant, breastfeeding, and/or planning to become pregnant and/or breastfeed during the study or within 30 days following the end of study participation
* Patients who are unable to swallow capsules
* Treatment with any investigational product within 3 months (or at least 5 half-lives, whichever is longer) of Visit 1. Treatment with any investigational product other than those provided by AGN during study participation will be a protocol violation, and the patient will be terminated from this study
* Employee or immediate relative of an employee of Allergan (AGN), any of its affiliates or partners, or of the study center
* Patients or patients whose parent/guardian/ legally authorized representative (LAR) and/or caregivers are unable to speak and understand English (or their native language if this can be accommodated by the site and is approved by the Sponsor) sufficiently to understand the nature of the study, to provide informed assent/consent, or to allow the completion of all study assessments
* Unable or unlikely to comply with the study protocol or are unsuitable for any other reason, Other Criteriaas judged by the Investigator

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Radecki, PhD, Study Director — Allergan
Locations (51):
- United States (51):
  - Woodland International Research Group, Little Rock, Arkansas
  - Care Access Research, Beverly Hills, Beverly Hills, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Imperial, California
  - Alliance Research, Long Beach, California
  - Excell Research, Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Children's National Health System, Washington D.C., District of Columbia
  - Advanced Research Institute of Miami, Homestead, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Zynak Clinical, Lauderdale Lakes, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Attalla Consultants, LLC, Smyrna, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Inova Clinical trials and Research Center, Tyrone, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR Conventions Limited, Naperville, Illinois
  - AMR-Baber Research, Inc., Naperville, Illinois
  - KU Wichita Clinical Trial Unit, Wichita, Kansas
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Millennium Center for Clinical Research, Creve Coeur, Missouri
  - Millennium Psychiatric Associates, LLC, St Louis, Missouri
  - Alivation Research, Lincoln, Nebraska
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Finger Lake Clinical Research, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Department of Psychiatry, Columbus, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - CincyScience, West Chester, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - BioBehavioral Research of Austin, Austin, Texas
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Roque Medical Trails LLC, Dallas, Texas
  - El Campo Clinical Trials, El Campo, Texas
  - Mech Healthcare Associates, Frisco, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Northpointe Psychiatry, Lewisville, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - AIM Trials, Plano, Texas
  - Clinical Trials of Texas, Inc. (CTT), San Antonio, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Radecki DT, Robieson WZ, Gopalkrishnan M, Greenberg E, Aziz M. Safety and Efficacy of Levomilnacipran Extended Release in Pediatric Patients Aged 7-17 Years with Major Depressive Disorder: Results of Two Phase 3, Randomized, Double-Blind Studies. J Child Adolesc Psychopharmacol. 2024 Jun;34(5):241-250. doi: 10.1089/cap.2023.0080. Epub 2024 May 3. PMID 38700708

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Treatment Period (8 Weeks)
Arm/Group | Placebo | Levomilnacipran ER 40-80 mg/Day | Fluoxetine 20 mg/Day
Started | 164 | 169 | 168
Safety Population (Safety Population included all participants in the Randomized Population (all participants who underwent a Screening Visit, received a screening number, for whom informed consent was obtained, and who were randomized to a treatment group in the study) who received at least 1 dose of double-blind investigational product.) | 160 | 166 | 166
Completed | 146 | 146 | 144
Not Completed | 18 | 23 | 24
Not completed — Adverse Event | 1 | 2 | 5
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 10 | 9
Not completed — Lost to Follow-up | 7 | 7 | 6
Not completed — Protocol Deviation | 1 | 1 | 1
Not completed — Non-compliance with Study Drug | 1 | 1 | 1
Not completed — Reason not Specified | 1 | 1 | 2
Period: Double-blind Down-taper Period (1 Week)
Arm/Group | Placebo | Levomilnacipran ER 40-80 mg/Day | Fluoxetine 20 mg/Day
Started | 140 | 141 | 140
Completed | 140 | 139 | 138
Not Completed | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants in the Randomized Population who received at least 1 dose of double-blind investigational product.
Groups:
- Levomilnacipran ER 40-80 mg/Day: Levomilnacipran ER capsules, orally, 10 mg/day on Days 1 to 3, 20 mg/day on Days 4 to 7, and 40 mg/day from Week 2 through Week 8 of the Double-blind Treatment Period followed by levomilnacipran ER 40 mg/day on Days 1 and 2, and then 20 mg/day from Day 3 through Day 7 in the Down-taper Period. Based on therapeutic response and tolerability, an additional dose increase to 80 mg/day was permitted at Week 3 of the Double-blind Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Levomilnacipran ER 40-80 mg/Day | Fluoxetine 20 mg/Day | Total
Number analyzed (Participants) | 160 | 166 | 166 | 492
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (2.48) | 13.7 (2.56) | 13.3 (2.66) | 13.5 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 99 | 105 | 318
  Male | 46 | 67 | 61 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 40 | 40 | 125
  Not Hispanic or Latino | 115 | 126 | 126 | 367
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 2 | 4 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 54 | 61 | 58 | 173
  White | 102 | 96 | 104 | 302
  More than one race | 1 | 5 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Children's Depression Rating Scale-Revised (CDRS-R) Total Score [Mean (Standard Deviation); unit: score on a scale] — The CDRS-R is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6-17 years. It contains 17 ordinally-scaled items that evaluate the presence and severity of symptoms commonly associated with childhood depression and is scored on a 1-to-5- or 1-to-7-point scale. Rating of 1 indicates normal function. The CDRS-R total score ranges from 17 to 113; higher scores indicate more severe depression. Population: Intent-to-Treat (ITT) Population included all participants in the Safety Population who had the Baseline and at least 1 post-baseline assessment of the CDRS-R total score. If a participant received an intervention different from the planned intervention, the participant is counted in the planned group.
  score on a scale
    number analyzed (Participants) | 159 | 162 | 166 | 487
    (all) | 60.8 (8.99) | 60.8 (9.17) | 60.9 (9.88) | 60.8 (9.34)
Clinical Global Impression-Severity (CGI-S) Scale [Mean (Standard Deviation); unit: score on a scale] — The CGI-S is a clinician-rated scale used to rate the severity of the participant's current state of mental illness compared with major depressive disorder (MDD) population. The participant was rated on a scale from 1 to 7, where 1=normal, not at all ill and 7=among the most extremely ill participants. Higher score indicates worsening of mental illness. Population: ITT Population included all participants in the Safety Population who had the Baseline and at least 1 post-baseline assessment of the CDRS-R total score. If a participant received an intervention different from the planned intervention, the participant is counted in the planned group.
  score on a scale
    number analyzed (Participants) | 159 | 162 | 166 | 487
    (all) | 4.8 (0.64) | 4.7 (0.64) | 4.8 (0.60) | 4.8 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Children's Depression Rating Scale- Revised (CDRS-R)
Description: The CDRS-R is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6-17 years. It contains 17 ordinally-scaled items that evaluate the presence and severity of symptoms commonly associated with childhood depression and is scored on a 1-to-5- or 1-to-7-point scale. Rating of 1 indicates normal function. The CDRS-R total score ranges from 17 to 113; higher score indicates more severe depression. A negative change from Baseline indicates improvement. Mixed Model for Repeated Measures (MMRM) was used for analysis.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT Population included all participants in the Safety Population who had the baseline and at least 1 postbaseline assessment of the CDRS-R total score. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Levomilnacipran ER 40-80 mg/Day | Fluoxetine 20 mg/Day
Number analyzed (Participants) | 146 | 148 | 144
score on a scale | -21.3 (1.01) | -23.0 (1.01) | -23.1 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER 40-80 mg/Day; Test type: Superiority; p = 0.2215, Mixed Model for Repeated Measures; Least Square Mean Difference = -1.7, 95% CI 2-sided [-4.49 to 1.04], Standard Error of Mean 1.41 — Estimates and p-values are based on MMRM with treatment group, pooled study center, visit, and treatment group-by-visit interaction as fixed effects, and Baseline and Baseline-by-visit as covariates using an unstructured covariance matrix
Statistical Analysis 2: Comparison: Placebo vs Fluoxetine 20 mg/Day; Test type: Superiority; p = 0.1964, Mixed Model for Repeated Measures; Least Square Mean Difference = -1.8, 95% CI 2-sided [-4.59 to 0.95], Standard Error of Mean 1.41 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scale
Description: The CGI-S is a clinician-rated scale used to rate the severity of the participant's current state of mental illness compared with MDD population. The participant was rated on a scale from 1 to 7, where 1=normal, not at all ill and 7=among the most extremely ill participants. Higher score indicates worsening of mental illness. A negative change from Baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT Population included all participants in the Safety Population who had the Baseline and at least 1 post-baseline assessment of the Children's Depression Rating Scale-Revised (CDRS-R) total score. If a participant received an intervention different from the planned intervention, the participant is counted in the planned group. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Levomilnacipran ER 40-80 mg/Day | Fluoxetine 20 mg/Day
Number analyzed (Participants) | 146 | 148 | 144
score on a scale | -1.5 (0.10) | -1.6 (0.10) | -1.7 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER 40-80 mg/Day; Test type: Superiority; p = 0.6789, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.1, 95% CI 2-sided [-0.32 to 0.21], Standard Error of Mean 0.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Fluoxetine 20 mg/Day; Test type: Superiority; p = 0.1126, Mixed Model for Repeated Measures; Least Square Mean Difference = -0.2, 95% CI 2-sided [-0.48 to 0.05], Standard Error of Mean 0.13

ADVERSE EVENTS:
Time Frame: Up to approximately 9 weeks
Description: All-cause Mortality: All enrolled participants. Adverse Events: Safety Population included all participants in the Randomized Population who received at least 1 dose of double-blind investigational product. Data was collected and reported separately for the Double-blind Treatment Period and the Double-blind Down-taper Period.
Groups:
- Placebo (Double-blind Treatment Period): Matching placebo capsules once daily through 8 weeks in the Double-blind Treatment Period.
- Levomilnacipran ER 40-80 mg/Day (Double-blind Treatment Period): Levomilnacipran ER capsules, orally, 10 mg/day on Days 1 to 3, 20 mg/day on Days 4 to 7, and 40 mg/day from Week 2 through Week 8 of the Double-blind Treatment Period. Based on therapeutic response and tolerability, an additional dose increase to 80 mg/day was permitted at Week 3 of the Double-blind Treatment Period.
- Fluoxetine 20 mg/Day (Double-blind Treatment Period): Fluoxetine capsule, orally, 10 mg/day at Week 1, and 20 mg/day from Week 2 through Week 8 of the Double-blind Treatment Period.
- Placebo (Down-taper Period): Matching placebo capsules once daily on Days 1 through 7 in the Down-taper Period.
- Levomilnacipran ER 40-80 mg/Day (Down-taper Period): Levomilnacipran ER capsules, orally, 40 mg/day on Days 1 and 2, and then 20 mg/day from Day 3 through Day 7 in the Down-taper Period. Based on therapeutic response and tolerability, an additional dose increase to 80 mg/day was permitted at Week 3 of the Double-blind Treatment Period.
- Fluoxetine 20 mg/Day (Down-taper Period): Fluoxetine capsule, orally, 10 mg/day from Day 1 through Day 7 of the Down-taper Period.
Arm/Group | Placebo (Double-blind Treatment Period) | Levomilnacipran ER 40-80 mg/Day (Double-blind Treatment Period) | Fluoxetine 20 mg/Day (Double-blind Treatment Period) | Placebo (Down-taper Period) | Levomilnacipran ER 40-80 mg/Day (Down-taper Period) | Fluoxetine 20 mg/Day (Down-taper Period)
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/169 | 0/168 | 0/160 | 0/166 | 0/166
Serious Adverse Events (participants affected / at risk) | 1/160 | 1/166 | 4/166 | 1/160 | 0/166 | 0/166
Other Adverse Events (participants affected / at risk) | 32/160 | 44/166 | 37/166 | 3/160 | 3/166 | 1/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Treatment Period) (N=160) | Levomilnacipran ER 40-80 mg/Day (Double-blind Treatment Period) (N=166) | Fluoxetine 20 mg/Day (Double-blind Treatment Period) (N=166) | Placebo (Down-taper Period) (N=160) | Levomilnacipran ER 40-80 mg/Day (Down-taper Period) (N=166) | Fluoxetine 20 mg/Day (Down-taper Period) (N=166)
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Treatment Period) (N=160) | Levomilnacipran ER 40-80 mg/Day (Double-blind Treatment Period) (N=166) | Fluoxetine 20 mg/Day (Double-blind Treatment Period) (N=166) | Placebo (Down-taper Period) (N=160) | Levomilnacipran ER 40-80 mg/Day (Down-taper Period) (N=166) | Fluoxetine 20 mg/Day (Down-taper Period) (N=166)
Tachycardia (Cardiac disorders) | 0 | 10 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 16 | 5 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 11 | 12 | 0 | 0 | 0
Headache (Nervous system disorders) | 19 | 21 | 19 | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 9 | 2 | 5 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03569475/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT03569475/SAP_001.pdf